CLINICAL TRIAL: NCT05316792
Title: Evaluation of Femoral Cartilage Thickness After Treadmill and Tartan Track Walking in Healthy Individuals and Patients With Knee Osteoarthritis
Brief Title: Evaluation of Femoral Cartilage Thickness After Treadmill and Tartan Track Walking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PamukkaleU-Simsek-002
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Cartilage; Ultrasonography
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Case-Control Study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- knee osteoarthritis (Active Comparator): In patients with knee osteoarthritis, the thickness of the femoral articular cartilage will be measured with portable USG before and immediately after walking.
  Interventions: Other: walking
- healthy volunteers (Active Comparator): Femoral articular cartilage thickness will be measured with portable USG before and immediately after walking in healthy volunteers.
  Interventions: Other: walking

INTERVENTIONS:
Other: walking — 30 min walking on the treadmill and tartan floor

SUMMARY:
The aim of this study is to measure and compare the femoral cartilage deformation after walking on the treadmill and tartan floor in patients with knee osteoarthritis (OA) and healthy volunteers.

DETAILED DESCRIPTION:
The investigators will recruit 30 patients who will be applied to Physical Medicine and Rehabilitation outpatient clinic and diagnosed with knee OA according to American College of Rheumatology (ACR) criteria and 30 healthy volunteers matched for age and gender. The sociodemographic characteristics and detailed history of the patients included in the study will be questioned and recorded. After a detailed physical examination of all patients, weight and height will be measured, and body mass indexes (BMI) will be calculated. Participants' physical activity levels will be determined based on the World Health Organization's Global Physical Activity Questionnaire. This questionnaire has been reported to provide a valid and reliable estimate of physical activity, Turkish validity and reliability have been established.

A repeated measures design will be used in which healthy volunteers and patients with knee OA all complete all loading conditions (30min walking on the treadmill and tartan floor). For this, each group (healthy volunteers and knee OA patients) will first walk on the treadmill and then do tartan ground walking 1 week later. Femoral articular cartilage thickness before and immediately after walking will be measured with portable ultrasonography (USG) with a telemedicine feature.

Upon arrival at the treatment unit or area of the tartan track, participants will sit on a treatment table with their knees fully extended for 30 minutes to minimize the effects of previous activity on cartilage. All sessions will be completed at the same time of day to reduce daily variations in cartilage thickness. The dominant leg will be defined as the self-reported limb that the participant chooses to use to kick a ball. All post-load USG procedures will be achieved within 5 minutes after the loading condition. 3 images will be taken from each participant.

Two separate evaluators will measure to determine the reliability among the measurers.

To equalize the loading, the speed at which each participant walks on the treadmill in 30 minutes will be determined by the pedometer as a brisk walking speed (5 km/h). Again, each participant will walk on the tartan floor with a pedometer and walk for 30 minutes at an equal distance at the same pace as on the treadmill. The pedometer will give a warning when it is below or above the desired speed.

ELIGIBILITY:
Inclusion Criteria:

* Be over 40 years old
* Having been diagnosed with knee OA according to the ACR diagnostic criteria
* Being diagnosed with stage 1-2 knee OA according to the Kellgren-Lawrence staging criteria

Exclusion Criteria:

* Having a musculoskeletal or systemic disease that will prevent the exercise
* History or symptoms of lower extremity surgery, ligament injury, balance disorder, lower extremity injury in the last 6 months
* Presence of psychiatric or neurological disease affecting cooperation, cognitive and neurological functions

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic Evaluation | just before walking
  Femoral joint cartilage thickness will be measured with portable USG with telemedicine feature.
Ultrasonographic Evaluation | within 5 minutes after loading condition
  Femoral joint cartilage thickness will be measured with portable USG with telemedicine feature.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Alkan, Prof., Study Director — Pamukkale University